CLINICAL TRIAL: NCT07116993
Title: Comparative Effects of Ultrasound and Infrared on Pain, Range of Motion and Joint Health in Knee, Elbow and Ankle Joints in Patients With Hemophilia A: a Randomized Clinical Trial
Brief Title: Effects of Ultrasound and Infrared on Joint Pain and Movement in Hemophilia A Patients.
Acronym: Hemophilia A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danyal Ahmad (Other)
Responsible Party: Sponsor-Investigator, Danyal Ahmad, head supervior, University of Management and Technology Sialkot Pakistan
Organization: University of Management and Technology Sialkot Pakistan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: kuhs/dpt/umt-skt-017
Record Dates: First submitted 2024-10-30; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Hemophilia A
Keywords: hemophilia A; ultrasound; infrared; joint health
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ultrasound (Experimental): ultrasound group containing 15 participants who were given ultrasound therapy for 10 minutes along with the conventional physiotherapy.
  Interventions: Device: theraputic ultrasound
- infrared radiation (Experimental): infrared radiation group containing 15 participants who were treated with infrared therapy for 10 minutes along with the conventional physiotherapy.
  Interventions: Device: infrared radiation

INTERVENTIONS:
Device: theraputic ultrasound — Ultrasound is a mechanical sound wave with frequencies above human hearing, requiring a medium like air or tissue to travel, commonly used in imaging.
  Arms: ultrasound
Device: infrared radiation — Infrared, in contrast, is electromagnetic radiation associated with heat, doesn't need a medium, and is used in applications like thermal imaging and remote controls.
  Arms: infrared radiation

SUMMARY:
The study aims to compare the effectiveness of therapeutic ultrasound and infrared in managing hemarthrosis in patients with Hemophilia A, focusing on specific outcomes like joint pain, swelling, muscle atrophy, and range of motion.The main question to it is either one from both of the modalities are effective for hemophilia patients or not? comparison will be done to check the effectiveness of ultrasound and infrared on patients of both groups.

participants will:

1. get the treatment according to their respective groups
2. Both groups were given 4 sessions for 4 weeks.

DETAILED DESCRIPTION:
The data collection was started by the consent of the participants through the consent form. Then we randomly divided the patients into Group A and Group B. Group A participants were given Ultrasound therapy for 10 minutes with intensity of 1.5 W/m2 along with the conventional physiotherapy as well as home plan. Group B participants were given Infrared therapy for 10 minutes with moderate intensity along with the conventional physiotherapy as well as home plan. Both groups were given 4 sessions for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hemophilia A (Eid & Aly, 2015) .
2. Who had the Bleeding frequency of atleast once per week (Eid & Aly, 2015).
3. Males with hemophilia A
4. Irrespective of their therapeutic regime administered by their hematologists (Donoso-Úbeda, Meroño-Gallut, López-Pina, & Cuesta Barriuso, 2020) .

Exclusion Criteria:

1. Patients who had surgical procedures (Eid & Aly, 2015) .
2. Patients who were suffering from co-morbidities along with Hemophilia A.
3. Patients who had any other disability/deformity.
4. Who were receiving other physiotherapy treatment (Donoso-Úbeda et al., 2020) .
5. Who failed to sign the informed consent (Donoso-Úbeda et al., 2020)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — males with hemophilia A
Enrollment: 30 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
joint pain | 3 weeks
  Joint Pain: Measured using the Numerical Pain Rating Scale (NPRS) to quantify changes in pain severity. 0 indicates no pain while 10 indicates severe pain
ROM | 3 weeks
  Range of Motion (ROM): Measured using a goniometer to assess improvements in flexion and extension angles, measured in degrees, in the joint.
Swelling | 3 weeks
  Assessed based on circumference measurements around knee, elbow and ankle joint using inelastic tape measure in centimeters around the affected joint to detect reductions in swelling.

CONTACTS AND LOCATIONS:
Locations (1):
- Danyal Ahmad, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No